CLINICAL TRIAL: NCT03280173
Title: A Phase 1, Open-label, Randomized, Four-period, Four-sequence, Single-dose, Crossover Study In Healthy Volunteers, To Determine The Relative Bioavailability Of Pf-06291826 61 Mga Tafamidis Free Acid Soft Gelatin Capsules Compared To Commercial 4 × 20 Mg Tafamidis Meglumine Soft Gelatin Capsules Administered Under Fasted And Fed Conditions And The Effect Of Food On The Oral Bioavailability Of Pf-06291826 61 Mga Tafamidis Free Acid Soft Gelatin Capsules
Brief Title: A Study Comparing the Amounts of 2 Different Forms of Tafamidis (PF06291826), Both With and Without Food, In the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461054; 2017-002769-23 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 61 mgA tafamidis free acid soft gelatin capsule fed (Experimental): fasted
  Interventions: Drug: tafamidis
- 61 mgA tafamidis free acid soft gelatin capsule fasted (Experimental): fed
  Interventions: Drug: tafamidis
- 4 × 20 mg tafamidis meglumine soft gelatin capsules fed (Experimental): fed
  Interventions: Drug: tafamidis
- 4 × 20 mg tafamidis meglumine soft gelatin capsules fasted (Experimental): fasted
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — bioavailability study

SUMMARY:
2 different formulations of tafamidis will be compared under both fed and fasted conditions. Subjects will be fasted overnight or fed. After swallowing one of the tafamidis formulations, tafamidis blood concentrations will be measured periodically for 8 days. After 16 days, subjects will take a different formulation in the fed or fasted state or take the same formulation in the opposite feeding condition. This will be repeated, 16 days apart, until all subjects have taken each formulation both fed and fasted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria:

* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve 0-72 hours (AUC72) | 72 hrs
maximum observed plasma concentration (Cmax) | 168 hrs

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 168 hrs
Mean residence time (MRT) | 168 hrs
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 168 hrs
Plasma Decay Half-Life (t1/2) | 168 hrs
Area under the curve from zero to infinity (AUCinf) | 168 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461054&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Four-period%2C+Four-sequence%2C+Single-dose%2C+Crossover+Study+In+Healthy+Volunteers%2C+To+Determine+The+Relative+Bioavailability+Of+Pf-06291826+61+Mga+Tafamidis+Free+Acid+Soft+Gelatin+Capsules+Compared+To+Commercial+4+%C3%97+20+Mg+Tafamidis+Meglumine+Soft+Gelatin+Capsules+Administered+Under+Fasted+And+Fed+Conditions+And+The+Effect+Of+Food+On+The+Oral+Bioavailability+Of+Pf-06291826+61+Mga+Tafamidis+Free+Acid+Soft+Gelatin+Capsules